CLINICAL TRIAL: NCT04414657
Title: Development of a SARS-CoV-2 Research Biobank and Databank
Brief Title: USZ BioResource COVID-19
Status: Terminated | Type: Observational
Why Stopped: sufficient patient number reached; flattening out of pandemic in Switzerland
Sponsor: Regina Grossmann (Other)
Responsible Party: Sponsor-Investigator, Regina Grossmann, Dr. med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: CTC HFV2
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection; Biological Specimen Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMCs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sampling for biobank — blood sampling for biobank

SUMMARY:
Mono-centric. Blood sampling for biobank development, including linkage to patient data (resource for research on COVID19).

ELIGIBILITY:
Inclusion Criteria:

* m/f age > 18 years
* SARS-CoV-2 infektion (according to WHO guideline)
* hospitalisation, general ward
* acceptable language knowledge
* voluntary IFC and biobank appendix

Exclusion Criteria:

* contra indication for blood sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SARS-CoV-2 infektion (according to WHO guideline)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
blood sampling for biobank | 2 years
  development of a biobank

CONTACTS AND LOCATIONS:
Overall Officials: Regina Grossmann, Dr med, Study Director — Head of Clinical Trials Center University Hospital Zurich
Locations (1):
- University Hospital Zurich, Clinical Trials Center, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No